CLINICAL TRIAL: NCT01735045
Title: LSH Silicone Hydrogel Soft Hydrophilic Contact Lens for Daily Wear
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Szabocsik and Associates, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HF-2010-01
Record Dates: First submitted 2012-06-11; First posted 2012-11-28 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Group myopia control (Experimental): Subjects wearing contact lenses made of LSH (mangofilcon A) Soft (hydrophilic) Contact Lens for myopia control
  Interventions: Device: Lagado LSH (mangofilcon A) Soft (hydrophilic) Contact Lens
- Myopia Control (Active Comparator): Subjects wearing Benz 3GX (hioxifilcon B) Soft (hydrophilic) Contact Lens for myopia control
  Interventions: Device: Benz 3GX (hioxifilcon B) Soft (hydrophilic) Contact Lens

INTERVENTIONS:
Device: Lagado LSH (mangofilcon A) Soft (hydrophilic) Contact Lens — Daily Wear
  Arms: Test Group myopia control
Device: Benz 3GX (hioxifilcon B) Soft (hydrophilic) Contact Lens
  Arms: Myopia Control

SUMMARY:
This study is to evaluate the performance of the LSH (mangofilcon A) silicone hydrogel soft contact lenses when used as a daily wear contact lens for the correction of myopia.

ELIGIBILITY:
Inclusion Criteria:

* Have been advised that the contact lenses they will be wearing for the next 3 months are being used for investigational purposes and that their informed consent will be needed and documented prior to the start of the study.
* Visual acuity must be correctable to 20/30, with spherical lenses ranging in power from -1.00 to -5.00D, astigmatism≤1.50D.
* Have been successfully wearing soft (hydrophilic) contact lenses for at least one month prior to entering the study. (Success means both subject and practitioner are satisfied with visual acuity, comfort, and ocular physiology).
* Have non-diseased eyes which are normal or which have no preexisting ocular condition which would interfere with the patient's ability to adapt to the new pair of LSH Silicone Hydrogel Soft (hydrophilic) Contact Lenses. A normal eye is defined as one having all the following characteristics:

  1. No evidence of lid infection.
  2. No structural lid abnormality.
  3. No conjunctival abnormality or infection.
  4. A cornea which is clear with no edema, staining, vascularization or abnormal opacities, all as observed by slit lamp examination.
  5. No iritis.
  6. No other active ocular disease that would contraindicate use of the investigational lens.
  7. No GPC (giant papillary conjunctivitis, tarsal abnormality) Grade 2 or greater
* Use no ocular medication.
* Have no known sensitivity to solutions currently used for contact lens care.
* Have binocular correction with contact lenses.

Exclusion Criteria

* Astigmatism >1.50D
* No monocular or monovision fits may be included.
* Pregnant and lactating women are excluded from the study
* Minors (under age 18) are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Snelling Scale

SECONDARY OUTCOMES:
Slit Lamp Findings | 3 months
  Grading by the Slit Lamp Classification Scale

CONTACTS AND LOCATIONS:
Overall Officials: John M Szabocsik, PhD, Study Director
Locations (5):
- United States (5):
  - Glenda Secor, OD, Huntington Beach, California
  - Randall Sakamoto, Honolulu, Hawaii
  - Robert Davis, OD, Oak Lawn, Illinois
  - Douglas P. Benoit, OD, FAAO, Concord, New Hampshire
  - Stephen P. Byrnes, OD, FAAO, Londonderry, New Hampshire